CLINICAL TRIAL: NCT02120638
Title: Optimization of MDR-TB Treatment Regimen Based on the Molecular Drug Susceptibility Results of Pyrazinamide
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2013-260; 2013ZX10003008-003 (Other Grant/Funding Number: National Major Science and Technology Special Project)
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Multidrug Resistant Tuberculosis; Pyrazinamide
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Clinical Protocols; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyrazinamide Sensitive Comparator (Active Comparator): Pyrazinamide containing regimen: Regimen B1 - 6ZAmkLfxClrPto\6ZlfxClrPto
  * Six months of chemotherapy with Pyrazinamide,Amikacin,Levofloxacin,Clarithromycin,plus Prothionamide,followed by
  * Six months of Pyrazinamide,Levofloxacin,Clarithromycin,plus Prothionamide
  Interventions: Drug: Pyrazinamide containing regimen
- Pyrazinamide Resistant Comparator (Experimental): Regimen without Pyrazinamide: Regimen B2 - 6HAmkLfxClrPto\18HlfxClrPto
  * Six months of chemotherapy with Isoniazid,Amikacin,Levofloxacin,Clarithromycin,plus Prothionamide,followed by
  * Eighteen months of Isoniazid,Levofloxacin,Clarithromycin,plus Prothionamide
  Interventions: Drug: Regimen without Pyrazinamide

INTERVENTIONS:
Drug: Pyrazinamide containing regimen — Pyrazinamide 33-50kg 1000-1750 mg daily, 51-70kg 1750-2000 daily, >70kg 2000-2500mg daily Amikacin 600mg daily Levofloxacin 33-70kg 750 mg daily, >70kg 1000 mg daily Clarithromycin 33-50kg 500 mg daily, >50kg 1000 mg daily Prothionamide 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily All treatment is taken daily, for a duration of up to 12 months depending on treatment arm.
  Arms: Pyrazinamide Sensitive Comparator
Drug: Regimen without Pyrazinamide — Isoniazid 600mg daily Amikacin 600mg daily Levofloxacin 33-70kg 750 mg daily, >70kg 1000 mg daily Clarithromycin 33-50kg 500 mg daily, >50kg 1000 mg daily Prothionamide 33-50kg 500 mg daily, 51-70kg 750 daily, >70kg 1000 mg daily All treatment is taken daily, for a duration of up to 18 months depending on treatment arm.
  Arms: Pyrazinamide Resistant Comparator

SUMMARY:
Multidrug resistant tuberculosis (MDR-TB) is difficult to treat and raises a great challenge to TB control program. That pyrazinamide can shorten the course of treatment and facilitate bacilli clearance has been proved recently. In 2011, WHO recommended to use pyrazinamide throughout the course of treatment for MDR-TB. However, pyrazinamide susceptibility testing has not been widely used in clinic. And the conventional testing is time-consuming and unreliable. In contrast, the detection of pncA and rpsA mutations with molecular methods can provide rapid results of pyrazinamide susceptibility. The purpose of this study is to evaluate the efficacy of the introduce the molecular testing of pyrazinamide susceptibility in optimizing the MDR-TB treatment regimen.

DETAILED DESCRIPTION:
This is a phase 3, open labeled, prospective cohort study to evaluate the molecular testing of pyrazinamide susceptibility in optimizing the MDR-TB treatment regimen. Approximately 100 participants will be given the molecular detection of pncA and rpsA mutations and divide into to the pyrazinamide sensitive comparator group and the pyrazinamide resistant group based on the susceptibility results. For the pyrazinamide sensitive group, the regimen contains six months of chemotherapy with pyrazinamide, amikacin, levofloxacin, plus prothionamide, followed by six months of pyrazinamide, levofloxacin, clarithromycin, plus prothionamide. For the pyrazinamide resistant group, the regimen contains six months of chemotherapy with isoniazid, amikacin, levofloxacin, plus prothionamide, followed by eighteen months of isoniazid, levofloxacin, clarithromycin, plus prothionamide.

The participants will be followed up to 24 months after the start of the treatment. The primary outcome is the sputum culture conversion and the adverse events. Safety evaluations that will be performed are the routine lab tests, blood glucose, hearing , vital signs, ECG, reporting of adverse events, physical examinations and X-rays.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with active tuberculosis
* Patients who are smear positive and sputum culture positive for tuberculosis
* History of active tuberculosis less than 3 years
* With less than 2 times of previous antituberculous therapy
* The patients should be voluntarily entering the study and willing to sign up the consent form after full knowledge of the risks, schedule, drug features of this study.
* MDR-TB is defined as resistance to the following two drugs: Isoniazid and Rifampicin.
* Extensively drug-resistant(XDR-TB) is defined as resistance to any flouroquinolones and any one of the three second-line antituberculous injections (capreomycin, kanamycin, amikacin)
* The study enrolled MDR-TB subjects and excluded XDR-TB subjects. If MDR-TB subjects is also resistant to flouroquinolones or capreomycin( kanamycin, amikacin), the subjects is included in the study as pre-XDR TB patients.

Exclusion Criteria:

* Known allergy or intolerance to the drugs in this study
* Liver damage (Hepatic encephalopathy; ascites; prothrombin time prolonged 2 seconds compared with normal controls; blood bilirubin 3 times greater than the upper limit of the normal range)
* Platelets <150x109 / L, WBC < 3x109 / L.
* Abnormal ECG (Male patients with prolonged QT interval exceeding 430ms, Female patients with prolonged QT interval exceeding 450ms)
* Serum creatinine 1.5 times higher than upper limit
* Fasting blood-glucose higher than 8.0 mmol/L
* Patients who are on medication that effect the results of the drugs in this study
* Karnofsky score<50% (see appendix)
* Women who are pregnant or breastfeeding
* HIV positive
* Participating in other clinical trials in the past three months
* Patients with mental illness and severe neurosis
* Patients who have poor compliances
* Any special circumstances in which the research physicians believe that is not suitable for this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The Median Time to Sputum Culture Conversion | 24 months

SECONDARY OUTCOMES:
The Percentage of treatment success | 24 months
  Treatment success is defined as：
  1. During the last 12 months of treatment，participants have at least 5 sputum cultures negative taken at least 30 days apart.
  2. During the last 12 months of treatment，participants have only one sputum culture positive, followed by at least 3 consecutive sputum cultures negative taken at least 30 days apart, without symptoms progression.
  3. Participants complete the treatment, but less than 5 culture results are available.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, PhD, Principal Investigator — Huashan Hospital of Fudan University, Shanghai, China;Johns Hopkins University, Baltimore, Maryland, USA; Wenhong Zhang, PhD,MD, Principal Investigator — Huashan Hospital of Fudan University, Shanghai, China
Locations (11):
- China (11):
  - Chongqing Pulmonary Hospital, Chongqing, Chongqing Municipality
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Fifth People's Hospital of Wuxi, Wuxi, Jiangsu
  - Xinjiang Chest Hospital, Ürümqi, Xinjiang
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The Affiliated Hospital of Luzhou Medical College, Huzhou, Zhejiang
  - Wenling No.1 People's Hospital, Taizhou, Zhejiang
  - Ruian People's Hospital, Wenzhou, Zhejiang
  - Zhuji People's Hospital of Zhejiang Province, Zhuji, Zhejiang